CLINICAL TRIAL: NCT06718608
Title: Natural Evolution of Muscle Structure and Stiffness Following Brain Lesion
Acronym: Navomuss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024/31JUL/372
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Acute; Traumatic Brain Injury
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only one arm (Experimental)
  Interventions: Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: imaging — Magnetic resonance imaging (MRI) Shear wave elastography (SWE) Electronic oscillatory device (EOD)

SUMMARY:
We propose to carry out a single center, prospective, interventional trial to assess the natural evolution of lower limb muscle structure and muscle stiffness of hemiparetic patients following brain damage. Patients will be assessed two weeks, one month, three months and six months after their brain lesion.

Secondary objectives:

To compare the muscle stiffness and structure of patients who will develop muscle overactivity to patients who won't develop muscle overactivity.

To compare the muscle structure and muscle stiffness of the spastic lower limb muscles and the non-spastic lower limb muscles in the affected limb.

To compare the muscle structure and muscle stiffness of the affected and the non-affected lower limb.

To study the relationship between impairment and function by applying a comprehensive and original method to assess all aspects from muscle structure and mechanics to patient's functional capacities.

ELIGIBILITY:
Inclusion Criteria:

* Female or male ≥ 18 years and ≤ 80 years at screening
* Hemiparesis secondary to a first stroke or traumatic brain injury
* < 1 month post-stroke/brain injury Subjects must meet all of the inclusion criteria in order to be eligible to participate in the study.

Exclusion Criteria:

* Bilateral limb paresis
* Major cognitive impairments limiting the functional evaluation
* Neurological or orthopedic affection interfering with the paretic limbs function
* Underlying neuromuscular disease (e.g. myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis)
* Contraindication to perform MRI Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Muscle elasticity | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  Muscle elasticity measured by shear wave elastography, expressed in m/s. A smaller shearwave velocity indicates a better outcome

SECONDARY OUTCOMES:
muscle volume | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  muscle volume measured by magnetic resonance imaging, expressed in mm3. A greater muscle volume indicates a better outcome
muscle fat fraction | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  muscle fat fraction measured by magnetic resonance imagine, expressed in % . A smaller fat fraction indicates a better outcome

OTHER OUTCOMES:
passive range of motion | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  expressed in angles °. The greater the angle, the better the outcome
modified ashworth scale | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  minimum score:0; maximum score: 4. A higher score indicates a greater spasticity thus a worse outcome
modified Tardieu scale | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  minimum score:0; maximum score: 4. A higher score indicates a greater spasticity thus a wourse outcome
Fugl-meyer score (Lower extremity; motor function) | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  maximum score of 34. The highest the score, the better the motor function
10 meter walk test | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  Expressed in seconds. A reduced time indicates a better outcome
Timed Up And Go | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  Expressed in seconds. A reduced time indicates a better outcome
Berg balance scale | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  maximum score of 56. The highest the score, the better the balance
Abiloco | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  maximum score of 13. The highest the score, the better the outcome
Stroke Impact Scale | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  maximum score of 295. The highest the score, the better the outcome
Functional ambulation category | 2 weeks, 1 month, 3 months, 6 months after brain lesion
  maximum score of 5. The highest the score, the better the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gaetan Stoquart, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No